CLINICAL TRIAL: NCT02180854
Title: Correlation Between Monitoring Frequency and Clinical Deterioration in Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, John Asger Petersen, M.D., Consultant in Critical Care Medicine, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Delstudie4
Record Dates: First submitted 2014-06-27; First posted 2014-07-03 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: In-hospital Deterioration; Intra Hospital Cardiac Arrest; Sudden Death
Keywords: Early warning score; Rapid response systems; Medical emergency team
MeSH Terms: conditions — Death, Sudden | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (8 hours) (Experimental): EWS every 8 hours
  Interventions: Other: Increased monitoring frequency
- Control (12 hours) (Active Comparator): EWS every 12 hours
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group
  Arms: Control (12 hours)
Other: Increased monitoring frequency
  Arms: Intervention (8 hours)

SUMMARY:
Acute deterioration among hospitalised patient can result in serious adverse events like cardiac arrest, unexpected death or unanticipated intensive care unit (ICU) admission. Most events are preceeded by deteriorating vital signs, and potentially avoidable.

To detect and treat hospitalised at-risk patients early an early warning score (EWS) was introduced at the investigator site. EWS measures of a number of physiological parameters that are aggregated to a common score, that directs monitoring frequency, clinical interventions and competency of the provider.

Patients with low scores (0 - 1) are monitored every 12th hour and seldom experience serious adverse events. The optimal monitoring frequency for this group is unknown, and presently based on a compromise between patient safety and work load issues.

The aim of the present study is to explore if an 8 hourly monitoring interval (intervention) is correlated with a better outcome than 12 hour intervals (control), based on the number of patients that deteriorate to a higher EWS 24 hours after hospital admission in each group.

DETAILED DESCRIPTION:
Acute deterioration among hospitalised patient can result in serious adverse events like cardiac arrest, unexpected death or unanticipated intensive care unit (ICU) admission. Most events are preceeded by deteriorating vital signs, and potentially avoidable.

To detect and treat hospitalised patients at risk of clinical deterioration in a timely manner, an early warning score (EWS) was introduced at the investigator site. EWS includes measures for respiratory rate, arterial hemoglobin oxygen saturation, pulse rate, systolic blood pressure, level of consciousness according to AVPU score, temperature, and whether a patient receives supplementary oxygen. Each vital sign can be assigned between 0 to 3 points (supplementary oxygen 0 or 2) depending on how much it deviates from a predefined threshold; the values are added to an aggregated score from 0 to 20, higher scores indicating more severe disease. An escalation protocol that directs the type of clinical response and competency of the provider according to EWS triggers was also introduced as an integrated part of the system.

Patients with low scores (0 - 1) are monitored every 12th hour and seldom experience serious adverse events. The optimal monitoring frequency for this group is unknown, and presently based on a compromise between patient safety and work load issues.

The aim of the present study is to explore if an 8 hourly monitoring interval (intervention) is correlated with a better outcome than 12 hour intervals (control) in the group of patients that have an EWS of 0 or 1 on admission. Deterioration is based on the number of patients that deteriorate to a higher EWS 24 hours after the first EWS is measured. Since serious adverse events in this population are rare the primary outcome is clinical deterioration defined as number of patients with elevated EWS >/= 2 in each group, 24 hours after admission to the hospital.

This is a cluster-randomized, non-blinded, pragmatic, interventional study of acutely admitted, adult patients to surgical or medical wards at our hospital.

ELIGIBILITY:
Inclusion Criteria:

* first EWS on admission = 0 or 1
* age >/ = 18 years

Exclusion Criteria:

* chronically elevated EWS
* terminal disease and comfort care only
* conditions that warrant closer observation according to hospital guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with an EWS >/= 2 | 24 hours after first EWS after admission
  Clinical deterioration is correlated to elevated EWS

SECONDARY OUTCOMES:
Number of patients with an aggregated score of EWS >/= 5 or >/= 7 | 24 to 48 hours
EWS >/ = 2 | 48 hours
Mortality | 72 hours and 30 days
Length of hospital stay | 30 days
  Participants will be followed for the duration of their hospital stay, which is on average 3 - 5 days. Assessment of this data point will take place 30 days after admission.
Number of patients with an individual score of EWS >/= 3 | 24 to 48 hours after first EWS on admission
Number of serious adverse events during first 72 hours of admission | 72 hours
  Serious adverse events is either cardiac arrest, unexpected death or admission to intensive care unit (ICU)

OTHER OUTCOMES:
Number of EWS measurements performed during first 48 hours of admission | 48 hours
Number of MET calls during first 72 hours of admission | 72 hours
  MET = medical emergency team
Number of patients where escalation protocol is adhered to | 48 hours
  To evaluate whether hospital guidelines are followed in regard to:
  * monitoring frequency
  * review by physician (for EWS >/= 3)
  * review by MET or specialist (for EWS >/= 9)

CONTACTS AND LOCATIONS:
Overall Officials: John A Petersen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark